CLINICAL TRIAL: NCT03487757
Title: "The Effect of Core Stabilization Exercises on Respiratory Muscle Strength, Respiratory Functions and Postural Control in Hearing Impaired Children"
Brief Title: "Core Stabilization Exercises in Hearing Impaired Children"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Lecturer, PT, MSc, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvudtuncer01
Record Dates: First submitted 2018-03-28; First posted 2018-04-04 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hearing Disorders in Children; Core Stabilization; Respiratory Muscle Strength; Respiratory Functions; Postural Control

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): After recording the demographic and clinical information at the beginning of the study and after 8 weeks, respiratory muscle strength, respiratory functions and postural control evaluations will be performed to the children. They won't receive any intervention by this time. At the end of 8 weeks, they may be included in the 8-week physiotherapy program, which will be once a week and 45-60 minutes by supervision of physiotherapist and 4 days a week home exercise program. The program will include core stabilization exercise training.
  Interventions: Other: No Intervention
- Training Group (Experimental): After recording the demographic and clinical information at the beginning of the study, respiratory muscle strength, respiratory functions and postural control evaluations will be performed to the children. They will be included in the 8-week physiotherapy program, which will be once a week and 45-60 minutes by supervision of physiotherapist and 4 days a week home exercise program. The program will include core stabilization exercise training. After the eight week training program the evaluations will be repeated.
  Interventions: Other: Core Stabilization Exercises

INTERVENTIONS:
Other: Core Stabilization Exercises — Jeffrey's core stabilization exercise training protocol will be performed to the training group. This protocol includes exercises progressing gradually from level 1 to level 3. Level 1; static contraction training on a stable surface, level 2; dynamic training on a stable surface, level 3; dynamic and resistant training on an unstable surface.
  Arms: Training Group
Other: No Intervention — Since no training is given to the control group during the study period, it is ethically necessary to give the same training to the control group if the benefit is achieved when the study is completed.
  Arms: Control Group

SUMMARY:
In this study the investigators will examine the effects of core stabilization exercises on respiratory muscle strength, respiratory functions and postural control in hearing-impaired children.

DETAILED DESCRIPTION:
Hearing organs develop together with the vestibular system and work with close cooperation. Because of this close neuro-anatomic relationship; cochlear, semicircular canal, or both may cause damage to the vestibular dysfunction, resulting in imbalance. Sensory impairment in children with hearing loss may lead to decreased muscle strength and respiratory function with balance and coordination disorders. Core stabilization is provided anatomically with abdominal muscles at the front, spinal and gluteal muscles at the back, diaphragm at the top and pelvic floor and hip muscles at the bottom. Core stabilization training is a training to increase the strength, endurance and neuromuscular control of the aforementioned muscles.

When the literature is checked, the invetigators find that postural control is being evaluated in children with hearing impairment, but there are few studies evaluating respiratory functions. However, they did not encounter a study in which respiratory muscle strength was assessed in these children. In this study the investigators will examine the effects of core stabilization exercises on respiratory muscle strength, respiratory functions and postural control in hearing-impaired children.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-16
* Clinically diagnosed sensorineural hearing loss
* Prelingual hearing loss
* No neurological and orthopedic problems
* Absence of syndrome or disease that may lead to mental disorder, impaired development and impaired vision
* Not participating in any core stabilization, strengthening and balance program in the past six months
* No medication to affect respiratory functions in the past 3 months
* Parental permission for participation of child in the study

Exclusion Criteria:

* Intellectual disability for participating to the evaluation and training program
* Presence of chronic respiratory disease
* Not to join the training for more than 3 days

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | Eight weeks
  Change from baseline maximum inspiratory pressure and maximum expiratory pressure at 8 weeks

SECONDARY OUTCOMES:
Respiratory Functions-FVC | Eight weeks
  Change from baseline Forced Vital Capacity (FVC) at 8 weeks
Respiratory Functions-FEV1 | Eight weeks
  Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks
Respiratory Functions-PEF | Eight weeks
  Change from baseline Peak Expiratory Flow (PEF) at 8 weeks
Postural control-postural stability | Eight weeks
  Change from baseline postural stability test score in Biodex Balance System at 8 weeks
Postural control-limits of stability | Eight weeks
  Change from baseline limits of stability test score in Biodex Balance System at 8 weeks
Postural control-sensory integration | Eight weeks
  Change from baseline sensory integration and balance test core in Biodex Balance System at 8 weeks
Postural control-BESS | Eight weeks
  Change from baseline Balance Error Scoring System (BESS) test scores at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Tuncer D, Gurses HN. The Effects of Core Stabilization Exercises on Respiratory Muscle Strength, Respiratory Functions, and Postural Control in Children With Hearing Loss: A Randomized Controlled Trial. Ear Hear. 2024 Mar-Apr 01;45(2):306-315. doi: 10.1097/AUD.0000000000001428. Epub 2023 Oct 3. PMID 37784232